CLINICAL TRIAL: NCT02927080
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of ACE-083 in Patients With Facioscapulohumeral Muscular Dystrophy
Brief Title: Study of ACE-083 in Patients With Facioscapulohumeral Muscular Dystrophy (FSHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued as it did not achieve functional secondary endpoints.
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A083-02; ACE-083 (Other: Acceleron Pharma Inc.)
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150mg (Experimental): ACE-083 150 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200mg (Experimental): ACE-083 200 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200mg (Experimental): ACE-083 200 mg TA bilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg (Experimental): ACE-083 150 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg (Experimental): ACE-083 200 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg (Experimental): ACE-083 240 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- Placebo (Part 2, DB-PC) Tibialis Anterior (TA) (Placebo Comparator): Part 2, double-blind (DB) placebo-controlled (PC). Placebo TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
  Afterwards, participants were rolled over into the open-label portion and received ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083 or placebo
- ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg (Experimental): Part 2, double-blind placebo-controlled. ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
  Afterwards, participants were rolled over into the open-label portion and received ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083
- Placebo (Part 2, DB-PC) Biceps Brachii (BB) (Placebo Comparator): Part 2, double-blind placebo-controlled. Placebo BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
  Afterwards, participants were rolled over into the open-label portion and received ACE-083 240 mg Biceps Brachii (BB) bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083 or placebo
- ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg (Experimental): Part 2, double-blind placebo-controlled. ACE-083 240 mg Biceps Brachii (BB) bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
  Afterwards, participants were rolled over into the open-label portion and received ACE-083 240 mg Biceps Brachii (BB) bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
  Interventions: Drug: ACE-083

INTERVENTIONS:
Drug: ACE-083 — Recombinant fusion protein.
  Arms: ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150mg; ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg; ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200mg; ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg; ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200mg; ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg; ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg
Drug: ACE-083 or placebo — Recombinant fusion protein or normal saline.
  Arms: Placebo (Part 2, DB-PC) Biceps Brachii (BB); Placebo (Part 2, DB-PC) Tibialis Anterior (TA)

SUMMARY:
Study A083-02 is a multi-center, Phase 2 study to evaluate the safety, tolerability, pharmacodynamics (PD), efficacy, and pharmacokinetics (PK) of locally-acting ACE-083 in patients with Facioscapulohumeral muscular dystrophy (FSHD) to be conducted in two parts. Part 1 is open-label, dose-escalation and Part 2 is randomized, double-blind, and placebo-controlled.

DETAILED DESCRIPTION:
Part 1 (dose escalation, open-label) Part 1 will consist of up to 6 cohorts of patients and will evaluate multiple ascending dose levels of ACE-083 administered unilaterally or bilaterally to either the tibialis anterior (TA) or biceps brachii (BB) muscle(s). Patients in each cohort will be enrolled in a 4-week screening period before beginning treatment. A Safety Review Team (SRT) will meet to review data for each cohort when at least 4 patients within a cohort have completed their Day 43 visit prior to dose escalation of the next cohort. Study duration for Part 1 for each patient will be approximately 24 weeks, including a 4-week screening period, a 12-week treatment period, and an 8-week follow-up period after the last dose.

Part 2 (randomized, double-blind, placebo-controlled, with open-label extension) Prior to the initiation of Part 2, a review of safety and efficacy data from Part 1 will be conducted to determine whether cohorts for one or both muscles will be pursued in Part 2, as well as the recommended dose level for each muscle. A total of up to 56 new patients (28 patients per muscle) may be enrolled and randomized (1:1) to receive either ACE-083 (n=14/muscle) or placebo (n=14/muscle) bilaterally to either the TA or BB muscles (but not both). Patients will receive blinded study drug once every three weeks for approximately 6 months (9 doses).

Patients who complete the double-blind treatment period will immediately roll over to open-label treatment with ACE-083, receiving the same dose of active drug, bilaterally in either the TA or BB muscle, once every three weeks for approximately 6 months (8 doses). In Part 2, the SRT will periodically review blinded safety data for each muscle treated.

Study duration for Part 2 for each patient will be approximately 15 months, including a 1-month screening period, a 12-month treatment period (6-month double-blind, placebo-controlled and a 6-month open-label extension), and a 2-month follow-up period after the last dose

ELIGIBILITY:
Key Inclusion Criteria:

1. Age ≥ 18 years
2. Genetically confirmed Facioscapulohumeral muscular dystrophy type 1 (FSHD1) or FSHD2 (or a first-degree relative with genetically confirmed FSHD1 or FSHD2) and clinical findings meeting FSHD criteria
3. Part 1 TA cohorts:

   1. 6-minute walk distance (6MWD) ≥ 150 meters (without a brace)
   2. Mild to moderate weakness in left and/or right ankle dorsiflexion

   Part 1 BB cohorts:

   a. Mild to moderate weakness in left and/or right elbow flexion

   Part 2 TA cohorts:
   1. 6MWD ≥ 150 and ≤ 500 meters (without a brace)
   2. Mild to moderate weakness in left and right ankle dorsiflexion

   Part 2 BB cohorts:

   a. Mild to moderate weakness in left and/or right elbow flexion
4. Females of childbearing potential must have negative urine pregnancy test prior to enrollment and use highly effective birth control methods during study participation. Hormonal birth control use must be stable for at least 14 days prior to Day 1. Males must agree to use a condom during any sexual contact with females of childbearing potential while participating in the study even if he has undergone a successful vasectomy.

Key Exclusion Criteria:

1. Current/ active malignancy (e.g., remission less than 5 years duration), with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
2. Symptomatic cardiopulmonary disease, significant functional impairment, or other co morbidities that in the opinion of the investigator would limit a patient's ability to complete strength and/or functional assessments on study
3. Renal impairment (serum creatinine ≥ 2 times the upper limit of normal,(ULN))
4. Aspartate transaminase (AST) and/or alanine transaminase (ALT) ≥ 3 times ULN
5. Increased risk of bleeding (i.e., due to hemophilia, platelet disorders, or use of any anti-coagulation/platelet modifying therapies up to 2 weeks prior to Study Day 1; low dose aspirin [≤ 100 mg daily] is permitted)
6. Major surgery within 4 weeks prior to Study Day 1
7. Chronic systemic corticosteroids (≥ 2 weeks) within 4 weeks before Study Day 1 and for duration of study; intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids are permitted
8. Androgens or growth hormone within 6 months before Study Day 1 and for duration of study; topical physiologic androgen replacement is permitted
9. Any condition that would prevent MRI scanning or compromise the ability to obtain a clear and interpretable scan of the TA or BB muscles, as applicable (e.g., pacemaker, knee/hip replacement, or metallic implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (18):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hugo W. Moser Research Inst. at Kennedy Krieger Inc., Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester School of Medicine, Rochester, New York
  - Carolinas Healthcare System Neurosciences Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Montreal Neurological Institute & Hospital, Montreal, Quebec
- Spain (3):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario y Politécnico La Fe, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 22 November 2016, last subject completed 09 October 2019. The study was divided into parts; Part 1 was an open-label dose escalation study and had 6 cohorts and Part 2 was a randomized double-blind placebo controlled trial. Participants were recruited from 23 study centers in 3 countries (US, Canada and Spain).
Groups:
- ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) Unilateral: ACE-083 150 mg Tibialis Anterior (TA) unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) Unilateral: ACE-083 200 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) Bilateral: ACE-083 200 mg TA bilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) Unilateral: ACE-083 150 mg Biceps Brachii (BB) unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) Unilateral: ACE-083 200 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) Unilateral: ACE-083 240 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- Placebo (Part 2, DB-PC) Tibialis Anterior (TA): Double-Blind, Placebo-Controlled Placebo TA bilaterally, once every 3 weeks for up to 9 doses. Drug: Placebo Normal saline
- ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg: Double-Blind, Placebo-Controlled ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
- Placebo (Part 2, DB-PC) Biceps Brachii (BB): Double-Blind, Placebo-Controlled Placebo-BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
- ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg: Double-Blind, Placebo-Controlled ACE-083 240 mg BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
Period: Overall Study
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) Unilateral | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) Unilateral | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) Bilateral | ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) Unilateral | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) Unilateral | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) Unilateral | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Started | 6 | 6 | 6 | 6 | 7 | 6 | 15 | 14 | 15 | 14
Open-Label Extension From Part 2 Double Blind-Placebo Controlled (Patients who completed the double-blind (DB) treatment period continued into the open-label extension (OLE) period. Patients who received ACE-083 in the DB treatment period continued to receive the same dose of ACE-083 during the OLE period, and patients who received placebo during the DB treatment period were switched to receive ACE-083, 240 mg/muscle. In the OLE period, ACE-083 was administered bilaterally in either the TA or BB muscle once every 3 weeks for approximately 6 months (8 doses).) | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 13 | 14 | 12
Completed | 6 | 5 | 6 | 6 | 6 | 6 | 7 | 5 | 12 | 7
Not Completed | 0 | 1 | 0 | 0 | 1 | 0 | 8 | 9 | 3 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Not completed — Willingness to comply with protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 7 | 2 | 3
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population was used for the results posting for both parts of the study. The Safety Set consists of all patients who received at least one dose of the study drug (including placebo).
Groups:
- Placebo (Part 2, DB-PC) Tibialis Anterior (TA): Double-Blind, Placebo-Controlled Placebo- TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
- Placebo (Part 2, DB-PC) Biceps Brachii (BB): Double-Blind, Placebo-Controlled Placebo- BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
- ACE-083 (Part 2, DB-PC) Biceps Brachii (BB): Double-Blind, Placebo-Controlled ACE-083 240 mg BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
- Total: Total of all reporting groups
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150mg | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200mg | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200mg | ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 15 | 14 | 15 | 14 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 5 | 6 | 6 | 15 | 13 | 13 | 13 | 89
  >=65 years | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (4.3) | 43.7 (16.9) | 50.7 (7.6) | 52.2 (10.8) | 48.3 (17.6) | 41.2 (14) | 41.3 (14.5) | 50.9 (11.4) | 46.3 (17.2) | 46.7 (10.8) | 46.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 2 | 3 | 2 | 7 | 8 | 3 | 4 | 39
  Male | 3 | 3 | 2 | 4 | 4 | 4 | 8 | 6 | 12 | 10 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 5 | 6 | 6 | 7 | 5 | 14 | 14 | 14 | 14 | 91
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3
  White | 6 | 5 | 6 | 6 | 6 | 6 | 14 | 12 | 12 | 12 | 85
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 3 | 6 | 5 | 19
  United States | 6 | 5 | 4 | 6 | 7 | 5 | 9 | 7 | 6 | 8 | 63
  Spain | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 3 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability (Incidence of Adverse Events)
Description: The number of participants that had a least one Treatment Emergent Adverse Event for the duration of each of the respective study parts.
Time Frame: From initiation of treatment to Day 106 for Part 1 and Day 190 for Part 2
Population: The safety set population is all participants that received at least one dose of ACE-083 or placebo during the study.
Measure: Count of Participants; unit: Participants
Groups:
- ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150 mg: ACE-083 150 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200 mg: ACE-083 200 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein.
- ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200 mg: ACE-083 200 mg TA bilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- Placebo (Part 2, DB-PC) Tibialis Anterior (TA): Double-Blind, Placebo-Controlled Placebo-TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150 mg | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 15 | 14 | 15 | 14
Participants | 6 | 6 | 5 | 6 | 7 | 6 | 12 | 14 | 13 | 14

2. Primary Outcome: Safety and Tolerability (Severity of Adverse Events, Grade 3 or Higher).
Description: The number of participants that had a least one Treatment Emergent Adverse Event with CTCAE Grade 3 or Higher for the duration of each of the respective study parts.
Time Frame: From initiation of treatment to Day 106 for Part 1 and Day 190 for Part 2
Population: The safety set population is all participants that received at least one dose of ACE-083 or placebo during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150 mg | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 15 | 14 | 15 | 14
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

3. Primary Outcome: Safety and Tolerability (Severity of Adverse Events- Dose Interruption, Reduction and/or Drug Withdrawal)
Description: The number of participants that had a least one Treatment Emergent Adverse Event that led to dose interruption, dose reduction and/or drug withdrawn.
Time Frame: From initiation of treatment to Day 106 for Part 1 and Day 190 for Part 2
Population: The safety set population is all participants that received at least one dose of ACE-083 or placebo during the study.
Measure: Count of Participants; unit: Participants
Groups:
- ACE-083 (Part 1, Cohort 1b ) Biceps Brachii (BB) 150 mg: ACE-083 150 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150 mg | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 1b ) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7 | 6 | 15 | 14 | 15 | 14
Participants
  Dose interruption | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dose reduction | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Drug Withdrawal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

4. Primary Outcome: Total Muscle Volume (TMV) of the Treated Muscle in Patients With FSHD Administered ACE-083 or Placebo During Part 2 (Randomized, Controlled Portion)
Description: Total Muscle Volume (TMV)of the treated muscle in Patients with FSHD administered ACE-083 or placebo During Part 2 (randomized, controlled portion) from Baseline to Day 190. Total Muscle volume was measured by Magnetic Resonance Imaging (MRI). MRI was performed bilaterally on the tibialis anterior and the biceps brachii on Day 1, Day Day 43, Day 106, and Day 190. Baseline and Day 190 total muscle volume, means and standard deviations are reported.
Time Frame: Time Frame: From initiation of treatment to Study Visit Day 190
Population: The Per Protocol Set: All patients enrolled/randomized in the study who received at least one dose of the study drug (includes placebo) with no major protocol violations.
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 13 | 14 | 14
mm3
  Baseline Total Muscle Volume (TMV): number analyzed (Participants) | 14 | 13 | 13 | 14
  Baseline Total Muscle Volume (TMV) | 79708.77 (4507.67) | 85159.90 (22382.20) | 104788.87 (58681.86) | 89133.23 (48264.27)
  Day 190 Total Muscle Volume (TMV) | 81761.70 (43533.71) | 95739.04 (20689.98) | 109489.17 (56130.61) | 102131.94 (54608.84)

5. Primary Outcome: Percent Change of Total Muscle Volume (TMV) of the Treated Muscle in Patients With FSHD Administered ACE-083 or Placebo During Part 2 (Randomized, Controlled Portion)
Description: Percent Change of Total Muscle Volume (TMV)of the treated muscle in Patients with FSHD administered ACE-083 or placebo During Part 2 (randomized, controlled portion) from Baseline to Day 190. Total Muscle volume was measured by Magnetic Resonance Imaging (MRI). MRI was performed bilaterally on the tibialis anterior and the biceps brachii on Day 1, Day Day 43, Day 106, and Day 190. Percent Change from Baseline to Day 190 total muscle volume, mean and standard deviation is reported.
Time Frame: Time Frame: From initiation of treatment to Study Visit Day 190
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 13 | 14 | 14
percent change | 5.46 (7.32) | 14.20 (10.72) | 1.07 (8.08) | 20.41 (16.64)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; D190 Percent change from baseline in TMV; Test type: Superiority — Percent Change in Total Muscle Volume (TMV) of the TA muscle in patients with FSHD administered ACE-083 when compared to placebo During Part 2 (randomized, controlled portion); p = 0.0138, ANCOVA; Mean Difference (Net) = 9.54, 90% CI 2-sided [3.17 to 15.92], Standard Error of Mean 3.876
Statistical Analysis 2: Comparison: Placebo (Part 2, DB-PC) Biceps Brachii (BB) vs ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; D190 Percent change from baseline in TMV; Test type: Superiority — Percent Change in Total Muscle Volume (TMV) of the BB muscle in patients with FSHD administered ACE-083 when compared to placebo During Part 2 (randomized, controlled portion); p < 0.0001, ANCOVA; Mean Difference (Net) = 16.39, 90% CI 2-sided [9.75 to 23.02], Standard Error of Mean 4.032

6. Secondary Outcome: Percent Change in Total Muscle Volume (TMV) in Muscle in Patients With FSHD Administered ACE-083 During Part 1 (Open-label, Dose-escalation Portion)
Description: Percent Change in Total Muscle Volume (TMV) in muscle in patients with FSHD administered ACE-083 During 1 (open-label, dose-escalation portion) from Baseline to Day 106. Total Muscle volume was measured by Magnetic Resonance Imaging (MRI). MRI was performed bilaterally on the tibialis anterior and the biceps brachii on Day 1, Day Day 43, and Day 106, change from Baseline and Day 106 reported.
Time Frame: Time Frame: From initiation of treatment to Study Visit Day 106
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | ACE-083 (Part 1, Cohort 1a) Tibialis Anterior (TA) 150 mg | ACE-083 (Part 1, Cohort 2a) Tibialis Anterior (TA) 200mg | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) 200 mg | ACE-083 (Part 1, Cohort 1b) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
percent change | 8.1 (3.5) | 18.3 (3.7) | 19.7 (2.8) | 8.2 (6.0) | 17.1 (7.8) | 16.2 (4.7)

7. Secondary Outcome: Absolute Change in Fat Fraction (FF) of the Muscle in Patients With FSHD Administered ACE-083 or Placebo During Part 2 (Randomized, Controlled Portion)
Description: Absolute change in Fat Fraction (FF) of the muscle in patients with FSHD administered ACE-083 or Placebo During Part 2 (randomized, controlled portion) from Baseline to Day 190. Absolute change in intramuscular fat fraction in the tibialis anterior and biceps brachii were measured by Magnetic Resonance Imaging (MRI). MRI was performed bilaterally on the tibialis anterior and the biceps brachii on Day 1, Day Day 43, Day 106, and Day 190, change from Baseline and Day 190 reported.
Time Frame: Time Frame: From initiation of treatment to Study Visit Day 190
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo (Part 2, DB-PC) Bicpes Brachii (BB): Double-Blind, Placebo-Controlled Placebo- BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
Arm/Group | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Bicpes Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 13 | 14 | 14
Percent change | -0.32 (0.888) | -3.05 (0.946) | 1.03 (0.955) | -0.22 (0.978)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; D190 Absolute change from baseline in FF for the TA group administered ACE-083 when compared to Placebo in part 2; Test type: Superiority; p = 0.0359, ANCOVA; Mean Difference (Final Values) = -2.73, 90% CI 2-sided [-4.86 to -0.59], Standard Error of Mean 1.299
Statistical Analysis 2: Comparison: Placebo (Part 2, DB-PC) Bicpes Brachii (BB) vs ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; D190 Absolute change from baseline in FF for the BB group administered ACE-083 when compared to Placebo in part 2; Test type: Superiority; p = 0.3582, ANCOVA; Mean Difference (Final Values) = -1.25, 90% CI 2-sided [-3.49 to 0.99], Standard Error of Mean 1.359

8. Secondary Outcome: Percent Change From Baseline in Function of Tibialis Anterior, Part 2 (Randomized, Controlled Portion)
Description: Percent change from baseline in function of Tibialis Anterior during Part 2 assessed by: 6-minute walk test, 10 meter walk/run and 4-stair climb (ascend)
Time Frame: From initiation of treatment (Study Day 1) to Study Visit Day 190
Population: Per Protocol Set: All patients enrolled/randomized in the study who received at least one dose of the study drug (includes placebo) with no major protocol violations.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg
Number analyzed (Participants) | 14 | 13
percent change
  D190 6MWD from baseline | 8.56 (2.764) | 3.28 (2.937)
  D190 time to complete 10mW/R from baseline | -8.59 (3.351) | -3.90 (3.585)
  D190 4-stair ascend time from baseline | -5.20 (4.065) | -4.75 (4.318)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; D190 Percent change from baseline in 6 Minute Walk Test (MWT) distance from baseline; Test type: Superiority; p = 0.1945, ANCOVA; Mean Difference (Final Values) = -5.28, 90% CI 2-sided [-11.97 to 1.41], Standard Error of Mean 4.068
Statistical Analysis 2: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; D190 Percent change from baseline in time to complete a 10 meter walk/run; Test type: Superiority; p = 0.3451, ANCOVA; Mean Difference (Final Values) = 4.69, 90% CI 2-sided [-3.48 to 12.86], Standard Error of Mean 4.968
Statistical Analysis 3: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; D190 Percent change from baseline in time to complete 4-stair climb (ascend); Test type: Superiority; p = 0.9402, ANCOVA; Mean Difference (Final Values) = 0.45, 90% CI 2-sided [-9.47 to 10.37], Standard Error of Mean 6.030

9. Secondary Outcome: Percent Change From Baseline in Strength of Biceps Brachii, Part 2, Randomized-controlled
Description: Elbow flexion strength measured by hand-held dynamometry (quantitative muscle testing), maximum voluntary isometric contraction (MVIC).
Time Frame: From initiation of treatment (Study Day 1) to Study Visit Day 190
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 12
percent change | -3.54 (10) | 32.58 (10.44)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Biceps Brachii (BB) vs ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; Test type: Superiority; p = 0.0183, ANCOVA; Mean Difference (Final Values) = 36.12, 90% CI 2-sided [11.78 to 60.46], Standard Error of Mean 14.18

10. Secondary Outcome: Percent Change From Baseline in Performance of the Upper Limb (PUL) Mid-Level Elbow Dimension, Part 2, Randomized-controlled
Description: Percent Change from Baseline in Performance of the Upper Limb (PUL) Mid-Level Elbow Dimension, Part 2, Randomized-controlled, PUL from baseline to end of treatment (Day 190). The Performance of the Upper Limb is an assessment specifically designed for patients with Duchenne muscular dystrophy. The measures used in this study was a subset of the assessment. PUL was assessment by measures of high-level of movement (lifting weights of 50g, 200g, 500g and 1000g at shoulder height and above shoulder height) and mid-level movement by performing tasks with and without weights: hand to mouth with and without weights (50, 200g), hand to table, moving weights on table (100g, 200g, 500g and 1000g), lift light and heavy cans, stack light and heavy cans, remove lid from container, tearing paper).
Time Frame: From initiation of treatment (Study Day 1) to Study Visit Day 190
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 14
percent change | -1.19 (1.16) | 1.70 (1.17)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Biceps Brachii (BB) vs ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; Test type: Superiority; p = 0.0895, ANCOVA; Mean Difference (Final Values) = 2.89, 90% CI 2-sided [0.09 to 5.69], Standard Error of Mean 1.70

11. Secondary Outcome: Change From Baseline in Facioscapulohumeral Muscular Dystrophy-health Index (FSHD-HI), Patient-reported Outcome (PRO) Measures Part 2 (Randomized, Controlled Portion)- Total Score
Description: The facioscapulohumeral muscular dystrophy-health index (FSHD-HI) is a disease-specific patient-reported outcome (PRO) tool assessed by health-related quality of life and disease burden. The FSHD-HI questionnaire was designed to measure both overall FSHD health-related quality-of-life and 14 separate subdomains designed and based on patient interviews to measure total FSHD health-related quality-of-life, including both motor impairment and the social and emotional impact of FSHD. The 116 questions are combined into a total score, the score is transformed onto a percentage scale; with a range of 0-100, with 100 representing maximal disability, and lower scores representing decreasing disability, 0 representing no disability. The mean and standard deviation for baseline and day 190 are reported as is the absolute change from baseline to Day 190 during the randomized controlled portion of Part 2.
Time Frame: Time Frame: From initiation of treatment (Study Day 1) to Study Visit Day 190
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Biceps Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 14 | 13 | 14 | 14
score on a scale
  Baseline FSHD-HI total score | 37.65 (15.60) | 45.51 (28.44) | 45.52 (23.38) | 25.89 (21.78)
  Day 190 FSHD-HI total score | 39.44 (18.76) | 46.18 (29.15) | 47.27 (22.73) | 28.04 (27.31)
  Absolute Change Day 190 from Baseline | 1.79 (4.83) | 0.67 (6.02) | 1.75 (6.90) | 2.15 (12.76)
Statistical Analysis 1: Comparison: Placebo (Part 2, DB-PC) Tibialis Anterior (TA) vs ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg; Change from baseline in FSHD-HI, patient-reported outcome (PRO) measures Part 2 (Randomized, Controlled Portion)- Total Score for TA group part 2; compared to Placebo; Test type: Superiority; p = 0.5661, ANCOVA; Mean Difference (Final Values) = -1.98, 90% CI 2-sided [-7.67 to 3.70], Standard Error of Mean 3.459
Statistical Analysis 2: Comparison: Placebo (Part 2, DB-PC) Biceps Brachii (BB) vs ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg; Change from baseline in FSHD-HI, patient-reported outcome (PRO) measures Part 2 (Randomized, Controlled Portion)- Total Score for BB group part 2; compared to Placebo; Test type: Superiority; p = 0.9760, ANCOVA; Mean Difference (Final Values) = -0.11, 90% CI 2-sided [-6.06 to 5.84], Standard Error of Mean 3.618

12. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (200 mg Tibialis Anterior (TA) Bilaterally) Day 2, 24-hours After Dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration collection and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. Timepoints that have data are reported; Day 2, 24-hours after dose is reported.
Time Frame: Day 2, 24-hours after dose
Population: Pharmacokinetics Population: All patients who have received at least one dose of study drug and have sufficient pharmacokinetic (PK) samples collected and assayed for PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) Bilateral): ACE-083 200 mg TA bilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
Arm/Group | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) Bilateral)
Number analyzed (Participants) | 3
ng/mL | 42.03 (16.82)

13. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (200 mg Tibialis Anterior (TA) Bilaterally) Day 85, 6-hours After Dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. The timepoints for which data is available are reported. Day 86, 6-hours post-dose is reported.
Time Frame: Study Day 85 (6 hours post-dose)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACE-083 (Part 1, Cohort 3a) Tibialis Anterior (TA) Bilateral
Number analyzed (Participants) | 2
ng/mL | 63.9 (54.31)

14. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (200 mg Biceps Brachii (BB) Unilateral) Day 1, 6-hours Post-dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. The timepoints for which data is available are reported. Day 1, 6-hours post-dose, is reported.
Time Frame: Study Day 1, 6-hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) Unilateral
Number analyzed (Participants) | 3
ng/mL | 36.13 (12.7)

15. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (200 mg Biceps Brachii (BB) Unilateral) Day 85, 4-hours Post-dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. The timepoints for which data is available are reported.
Time Frame: Study Day 85, 4-hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACE-083 (Part 1, Cohort 2b) Biceps Brachii (BB) Unilateral
Number analyzed (Participants) | 3
ng/mL | 23.9 (2.87)

16. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (240 mg Tibialis Anterior (TA) Bilaterally) Day 2, 24- Hours Post-dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. The timepoints for which data is available are reported. Day 2, 24-hours post-dose is reported.
Time Frame: Day 2, 24-hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg Day 2, 24 Hours Post-dose: Double-Blind, Placebo-Controlled ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
Arm/Group | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg Day 2, 24 Hours Post-dose
Number analyzed (Participants) | 12
ng/mL | 65.08 (35.4)

17. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (240 mg Tibialis Anterior (TA) Bilaterally) Day 86, 24- Hours Post-dose
Description: Pharmacokinetic assessment included ACE-083 serum concentration and on a dosing day had a ±15 minute window for post-dose sample collection, based on the time of the first injection. The timepoints for which data is available are reported. Day 86, 24-hours post-dose is reported.
Time Frame: Day 86, 24-hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg
Number analyzed (Participants) | 11
ng/mL | 52.91 (37.74)

18. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (240 mg Biceps Brachii (BB) Bilaterally) Day 2, 24- Hours Post-dose
Description: as for outcome 16
Time Frame: Day 2, 24-hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg Day 1, 2 Hours Post-dose: Double-Blind, Placebo-Controlled ACE-083 240 mg BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
Arm/Group | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg Day 1, 2 Hours Post-dose
Number analyzed (Participants) | 14
ng/mL | 54.8 (20.97)

19. Secondary Outcome: ACE-083 Serum Concentration Following Local Intramuscular Administration (240 mg Biceps Brachii (BB) Bilaterally) Day 86, 24 Hours Post-dose
Description: as for outcome 17
Time Frame: Day 86, 24- hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg
Number analyzed (Participants) | 12
ng/mL | 46.87 (10.18)

ADVERSE EVENTS:
Time Frame: For part 1 (open-label; dose-escalation) the time frame is six months For part 2, there are two parts: randomized, double-blind, placebo-controlled and then an open-label portion- the total time frame for part 2 is fifteen months
Groups:
- ACE-083 (Part 1, Cohort 1a ) Tibialis Anterior (TA) 150mg: ACE-083 150 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 2a ) Tibialis Anterior (TA) 200mg: ACE-083 200 mg TA unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 3a ) Tibialis Anterior (TA) 200mg: ACE-083 200 mg TA bilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 2b ) Biceps Brachii (BB) 200 mg: ACE-083 200 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 1, Cohort 3b ) Biceps Brachii (BB) 240 mg: ACE-083 240 mg BB unilaterally, once every 3 weeks for up to 5 doses. Drug: ACE-083 Recombinant fusion protein.
- Placebo (Part 2, DB-PC) Bicpes Brachii (BB): Double-Blind, Placebo-Controlled Placebo BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: Placebo Normal saline
- ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg: ACE-083 240 mg BB bilaterally, once every 3 weeks for up to 9 doses.
  Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 2, Open-label) Tibialis Anterior (TA) 240 mg: ACE-083 240 mg TA bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
- ACE-083 (Part 2, Open-label) Biceps Brachii (BB) 240 mg: ACE-083 240 mg BB bilaterally, once every 3 weeks for up to 8 doses.
  Drug: ACE-083 Recombinant fusion protein
Arm/Group | ACE-083 (Part 1, Cohort 1a ) Tibialis Anterior (TA) 150mg | ACE-083 (Part 1, Cohort 2a ) Tibialis Anterior (TA) 200mg | ACE-083 (Part 1, Cohort 3a ) Tibialis Anterior (TA) 200mg | ACE-083 (Part 1, Cohort 1b ) Biceps Brachii (BB) 150 mg | ACE-083 (Part 1, Cohort 2b ) Biceps Brachii (BB) 200 mg | ACE-083 (Part 1, Cohort 3b ) Biceps Brachii (BB) 240 mg | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg | Placebo (Part 2, DB-PC) Bicpes Brachii (BB) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg | ACE-083 (Part 2, Open-label) Tibialis Anterior (TA) 240 mg | ACE-083 (Part 2, Open-label) Biceps Brachii (BB) 240 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/15 | 0/14 | 0/15 | 0/14 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/7 | 0/6 | 0/15 | 1/14 | 1/15 | 1/14 | 1/27 | 0/26
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 5/6 | 6/6 | 7/7 | 6/6 | 12/15 | 14/14 | 13/15 | 14/14 | 22/27 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACE-083 (Part 1, Cohort 1a ) Tibialis Anterior (TA) 150mg (N=6) | ACE-083 (Part 1, Cohort 2a ) Tibialis Anterior (TA) 200mg (N=6) | ACE-083 (Part 1, Cohort 3a ) Tibialis Anterior (TA) 200mg (N=6) | ACE-083 (Part 1, Cohort 1b ) Biceps Brachii (BB) 150 mg (N=6) | ACE-083 (Part 1, Cohort 2b ) Biceps Brachii (BB) 200 mg (N=7) | ACE-083 (Part 1, Cohort 3b ) Biceps Brachii (BB) 240 mg (N=6) | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) (N=15) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg (N=14) | Placebo (Part 2, DB-PC) Bicpes Brachii (BB) (N=15) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg (N=14) | ACE-083 (Part 2, Open-label) Tibialis Anterior (TA) 240 mg (N=27) | ACE-083 (Part 2, Open-label) Biceps Brachii (BB) 240 mg (N=26)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACE-083 (Part 1, Cohort 1a ) Tibialis Anterior (TA) 150mg (N=6) | ACE-083 (Part 1, Cohort 2a ) Tibialis Anterior (TA) 200mg (N=6) | ACE-083 (Part 1, Cohort 3a ) Tibialis Anterior (TA) 200mg (N=6) | ACE-083 (Part 1, Cohort 1b ) Biceps Brachii (BB) 150 mg (N=6) | ACE-083 (Part 1, Cohort 2b ) Biceps Brachii (BB) 200 mg (N=7) | ACE-083 (Part 1, Cohort 3b ) Biceps Brachii (BB) 240 mg (N=6) | Placebo (Part 2, DB-PC) Tibialis Anterior (TA) (N=15) | ACE-083 (Part 2, DB-PC) Tibialis Anterior (TA) 240 mg (N=14) | Placebo (Part 2, DB-PC) Bicpes Brachii (BB) (N=15) | ACE-083 (Part 2, DB-PC) Biceps Brachii (BB) 240 mg (N=14) | ACE-083 (Part 2, Open-label) Tibialis Anterior (TA) 240 mg (N=27) | ACE-083 (Part 2, Open-label) Biceps Brachii (BB) 240 mg (N=26)
Injection site pain (General disorders) | 5 | 4 | 3 | 1 | 4 | 3 | 4 | 5 | 6 | 6 | 6 | 7
Injection site discomfort (General disorders) | 1 | 1 | 3 | 5 | 0 | 2 | 1 | 3 | 4 | 2 | 3 | 3
Injection site erythema (General disorders) | 0 | 2 | 3 | 2 | 1 | 3 | 0 | 6 | 5 | 3 | 1 | 9
Injection site swelling (General disorders) | 0 | 3 | 2 | 1 | 2 | 2 | 0 | 2 | 0 | 3 | 1 | 6
Injection site bruising (General disorders) | 1 | 1 | 2 | 4 | 4 | 5 | 2 | 2 | 10 | 9 | 1 | 15
Injection site paraesthesia (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 6 | 1 | 2 | 1 | 4
Vessel puncture site bruise (General disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 5 | 0 | 0
Injection site hemorrhage (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Injection site warmth (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site discoloration (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Application site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Injection site papule (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site coldness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site hematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site hypoesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site dysaesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 4 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 2 | 0 | 4
Acne pustular (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Restless leg syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudofolliculitis barbae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myoglobin blood increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seborrheic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal septal operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02927080/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT02927080/SAP_000.pdf